CLINICAL TRIAL: NCT00872170
Title: Pilot of Oral Sildenafil for the Treatment of Pulmonary Hypertension in Thalassemia With Comparison to Controls
Brief Title: Sildenafil to Improve Exercise Capacity in People With Thalassemia and Pulmonary Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 638; U01HL065238 (NIH)
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-01

CONDITIONS: Thalassemia; Hypertension, Pulmonary
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Thalassemia; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Participants with thalassemia who have pulmonary hypertension will receive sildenafil for 12 weeks.
  Interventions: Drug: Sildenafil
- Control (No Intervention): Participants with thalassemia who do not have pulmonary hypertension will be part of a control group and will only be undergoing screening/baseline assessments.

INTERVENTIONS:
Drug: Sildenafil — Participants will receive sildenafil for 12 weeks with the following therapy:
  50 mg of oral sildenafil three times a day (TID) increased to 100 mg TID as tolerated in adults and children greater than 50 kg; 1 mg/kg sildenafil TID without dose escalation in children less than 50 kg
  Other Names: Revatio; Viagra
  Arms: Intervention

SUMMARY:
Thalassemia is an inherited blood disorder that can result in mild to severe anemia. Many people with thalassemia also have pulmonary hypertension, which is high blood pressure in the arteries in the lungs. This study will evaluate the safety and effectiveness of the medication sildenafil at reducing blood pressure in the lungs of people with thalassemia and pulmonary hypertension.

DETAILED DESCRIPTION:
Thalassemia is an inherited blood disorder in which the body makes an abnormal form of hemoglobin-the protein in red blood cells that carries oxygen. A potential complication of thalassemia is pulmonary hypertension, which is a condition characterized by abnormally high blood pressure in the arteries of the lungs. People with thalassemia who have pulmonary hypertension tend to experience more health complications, including shortness of breath and a reduced exercise capacity, than people with thalassemia who do not have pulmonary hypertension. Sildenafil is a medication that is used to treat pulmonary hypertension; however, it has not yet been studied in people with thalassemia. The purpose of this study is to evaluate the safety and effectiveness of sildenafil at reducing blood pressure in the lungs of people who have thalassemia and pulmonary hypertension. Study researchers will also further compare the differences between people with thalassemia who have pulmonary hypertension and those who do not have pulmonary hypertension.

This study will enroll people with thalassemia who have pulmonary hypertension and a control group of people with thalassemia who do not have pulmonary hypertension. People with thalassemia and pulmonary hypertension will attend a baseline study visit at which time they will undergo the following procedures: medical history and medical record review; physical exam; a 6-minute walk test, which will measure how far participants can walk in 6 minutes; an echocardiogram to obtain images of the heart; blood collection; and for females, a urine collection. Participants will then begin taking sildenafil three times a day for 12 weeks. At study visits at Weeks 2, 4, and 8, participants will undergo repeat baseline testing, and some participants will take part in an exhaled nitric oxide test. At Week 12, participants will also undergo lung function testing and a chest magnetic resonance imaging (MRI) procedure.

Participants in the control group will attend one to three study visits at baseline, which will include the same baseline study procedures listed above, plus lung function testing, a chest MRI, a chest computed tomography (CAT) scan, and exhaled nitric oxide testing. They will not receive any medication or have any further study visits.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Alpha, beta, or E-beta thalassemia confirmed by hemoglobin (Hb)-electrophoresis or molecular diagnosis

Inclusion Criteria for Participants with Pulmonary Hypertension:

* Pulmonary hypertension, defined as a tricuspid regurgitant jet (TRjet) velocity by Doppler echocardiography greater than 2.5 m/s

Inclusion Criteria for Participants without Pulmonary Hypertension:

* Lack of pulmonary hypertension, defined as TRjet velocity by Doppler echocardiography less than 2.5 m/s

Exclusion Criteria:

* Pregnant or breastfeeding
* Hypersensitivity to arginine or sildenafil, based on prior use
* Any of the following medical conditions:

  1. Severe kidney insufficiency, defined as use of hemodialysis or serum creatinine at levels greater than 2.5 mg/dL at the time of screening
  2. Cardiac disease with adjustment of cardiac medications in the 60 days before study entry
  3. Symptomatic coronary artery disease, as indicated by a history of chest pain, angina, claudication, or surgery to treat coronary artery disease in the 1 year before study entry
  4. Stroke, defined as a new focal neurological deficit lasting more than 24 hours in the 45 days before study entry
  5. New diagnosis of pulmonary embolism by ventilation-perfusion scan, angiography, or any other technique in the 90 days before study entry
  6. History of retinal detachment or retinal hemorrhage in the 180 days before study entry
  7. Use of nitrate-based vasodilators, prostacyclin (inhaled, subcutaneous, or intravenous), endothelin antagonists, or any other medication for pulmonary hypertension
  8. Acute asthma exacerbation requiring use of prednisone in the 60 days before study entry
  9. Initiation or dosage increase of calcium channel blockers in the 30 days before study entry
  10. Initiation of any other cardiac or pulmonary medication in the 90 days before study entry
* Presence of any other condition, which in the opinion of the investigator, would make the person unsuitable for enrollment or could interfere with compliance in the study, including but not limited to alcohol or drug abuse
* No measurable TRjet on Doppler echocardiography (i.e., presence of pulmonary hypertension cannot be confirmed or ruled out)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Neufeld, MD, PhD, Principal Investigator — Boston Children's Hospital; Claudia Morris, MD, Study Chair — Children's Hospital and Research Institute Oakland; Charles Quinn, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Patricia Giardina, MD, Principal Investigator — Weill Medical College of Cornell; Janet Kwiatkowski, MD, Principal Investigator — Children's Hospital of Philadelphia; Nancy Olivieri, MD, Principal Investigator — Toronto General Hospital; John Porter, MD, Principal Investigator — University College, London; Ali Taher, MD, Principal Investigator — American University of Beirut Medical Center- Lebannon
Locations (1):
- Children's Hospital and Research Institute Oakland, Oakland, California, United States

REFERENCES:
- [Result] Morris CR, Kim HY, Wood J, Porter JB, Klings ES, Trachtenberg FL, Sweeters N, Olivieri NF, Kwiatkowski JL, Virzi L, Singer ST, Taher A, Neufeld EJ, Thompson AA, Sachdev V, Larkin S, Suh JH, Kuypers FA, Vichinsky EP; Thalassemia Clinical Research Network. Sildenafil therapy in thalassemia patients with Doppler-defined risk of pulmonary hypertension. Haematologica. 2013 Sep;98(9):1359-67. doi: 10.3324/haematol.2012.082065. Epub 2013 Apr 12. PMID 23585527

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Participants with thalassemia who have pulmonary hypertension received sildenafil for 12 weeks.
  Sildenafil : Participants received sildenafil for 12 weeks with the following therapy:
  50 mg of oral sildenafil three times a day (TID) increased to 100 mg TID as tolerated in adults and children greater than 50 kg; 1 mg/kg sildenafil TID without dose escalation in children less than 50 kg
- Control: Participants with thalassemia who do not have pulmonary hypertension were part of a control group and were only undergoing screening/baseline assessments.
Period: Overall Study
Arm/Group | Sildenafil | Control
Started | 14 | 13
Completed | 13 (One patient withdrew from study at week 2.) | 13
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All 27 patients (14 in the Sildenafil group and 13 in the control group) who completed the baseline visit were used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Control | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.3) | 33.7 (12.6) | 34.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10
  Canada | 2 | 2 | 4
  United Kingdom | 6 | 5 | 11
  Lebanon | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Six-minute Walk Test (6MWT) Distance From Baseline to Week 12 Among Sildenafil Group
Description: Change in six-minute walk test (6MWT) distance was calculated as 6MWT at week 12 minus 6MWT at baseline.
Time Frame: Baseline and Week 12
Population: Of 14 patients in the Sildenafil arm, 4 patients with discrepant Tricuspid Regurgitant Jet Velocity (TRV) measurements between the local site, core lab and NHLBI readings and 2 patients who had no 6MWT at 12 weeks were excluded. Patients in control group were only assessed at baseline. Therefore, 8 Sildenafil and 0 control patients were used.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Sildenafil
Number analyzed (Participants) | 8
meters | -1.38 (16.01)
Statistical Analysis 1: Comparison: Sildenafil; This study had 80% power at level alpha=0.05 to detect a 60 m change in 6MWT among N=10 participants, assuming a 60 m standard deviation for 12-week change; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

2. Secondary Outcome: Change in Tricuspid Regurgitant Jet Velocity (TRV) From Baseline to Week 12 Among Sildenafil Group
Description: Change in tricuspid regurgitant jet velocity (TRV) was calculated as TRV at week 12 minus TRV at baseline. The TRV provides an estimate of pulmonary artery pressure.
Time Frame: Baseline and Week 12
Population: Of 14 patients in the Sildenafil arm, 4 patients with discrepant Tricuspid Regurgitant Jet Velocity (TRV) measurements between the local site, core lab and NHLBI readings and one patient who withdrew from the study were excluded. Patients in control group were only assessed at baseline. Therefore, 9 Sildenafil and 0 control patients were used.
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
m/s | -0.45 (0.18)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

3. Secondary Outcome: Change in Echo Left Ventricular End Systolic Volume (LVESV) From Baseline to Week 12 Among Sildenafil Group
Description: Change in echo left ventricular end systolic volume (LVESV) was calculated as LVESV at week 12 minus LVESV at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ml
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
ml | -3.82 (0.98)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

4. Secondary Outcome: Change in Echo Left Ventricular End Diastolic Volume (LVEDV) From Baseline to Week 12 Among Sildenafil Group
Description: Change in echo left ventricular end diastolic volume (LVEDV) was calculated as LVEDV at week 12 minus LVEDV at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ml
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
ml | -7.89 (2.71)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

5. Secondary Outcome: Change in Plasma Arginine From Baseline to Week 12 Among Sildenafil Group
Description: Change in Plasma Arginine was calculated as Plasma Arginine at week 12 minus Plasma Arginine at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: µM
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
µM | 31.77 (15.81)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

6. Secondary Outcome: Change in Red Blood Cell (RBC) Arginine From Baseline to Week 12 Among Sildenafil Group
Description: Change in Red Blood Cell (RBC) Arginine was calculated as Red Blood Cell (RBC) Arginine at week 12 minus Red Blood Cell (RBC) Arginine at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: µM
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
µM | 3.67 (1.45)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

7. Secondary Outcome: Change in Soluble Platelet Selectin (sP-SELECTIN) From Baseline to Week 12 Among Sildenafil Group
Description: Change in Soluble platelet selectin (sP-SELECTIN) was calculated as sP-SELECTIN at week 12 minus sP-SELECTIN at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
ng/ml | 121.13 (57.56)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

8. Secondary Outcome: Change in Lactate Dehydrogenase (LDH) From Baseline to Week 12 Among Sildenafil Group
Description: Change in Lactate dehydrogenase (LDH) was calculated as LDH at week 12 minus LDH at baseline.
Time Frame: Baseline and Week 12
Population: Of 14 patients in the Sildenafil arm, 4 patients with discrepant Tricuspid Regurgitant Jet Velocity (TRV) measurements between the local site, core lab and NHLBI readings and 2 patients who had no LDH at 12 weeks were excluded. Patients in control group were only assessed at baseline. Therefore, 8 Sildenafil and 0 control patients were used.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Sildenafil
Number analyzed (Participants) | 8
U/L | 23.37 (35.98)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.33, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

9. Secondary Outcome: Change in Cell Free Hemoglobin From Baseline to Week 12 Among Sildenafil Group
Description: Change in Cell Free Hemoglobin was calculated as Cell Free Hemoglobin at week 12 minus Cell Free Hemoglobin at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ug/ml
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
ug/ml | -67.60 (48.03)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

10. Secondary Outcome: Change in Arginase Concentration From Baseline to Week 12 Among Sildenafil Group
Description: Change in Arginase concentration was calculated as Arginase concentration at week 12 minus Arginase concentration at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
ng/ml | -17.06 (16.25)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

11. Secondary Outcome: Change in Arginase Activity From Baseline to Week 12 Among Sildenafil Group
Description: Change in Arginase activity was calculated as Arginase activity at week 12 minus Arginase activity at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Sildenafil
Number analyzed (Participants) | 9
U/L | 0.33 (2.88)
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; p = 0.96, Mixed Models Analysis; Linear mixed models with participant-specific intercepts and slopes controlled for time effects were used

ADVERSE EVENTS:
Time Frame: up to Week 12
Description: At each follow-up visit, Sildenafil patients were interviewed for medical conditions, medical changes, and symptoms that have occurred since the last visit. An Adverse Event (AE) form was completed if any AE was reported. A Serious Adverse Event form was completed for all AEs rated as serious. No AEs were collected for the control group.
Arm/Group | Sildenafil | Control
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/0
Other Adverse Events (participants affected / at risk) | 11/14 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=14) | Control (N=0)
Vision/color disturbance (Eye disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=14) | Control (N=0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 0 (0)
Vision/color disturbance (Eye disorders) | 2 (3) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain-other: sciatic pain of left leg with associated back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INR increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Phlebitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Ocular/visual - other (shining outline on objects) (Eye disorders) | 1 (1) | 0 (0)
Prolonged erection (priapism) (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Of 14 patients in the Sildenafil arm, 4 patients with discrepant TRVs between the local site, core lab and NHLBI readings were excluded for the main analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes